CLINICAL TRIAL: NCT02705898
Title: Technology-Supported Physical Activity Intervention for Depressed Alcoholic Women
Brief Title: Lifestyle Physical Activity Intervention for Depressed Alcohol Dependent Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1507-001; R34AA024038 (NIH)
Record Dates: First submitted 2016-02-29; First posted 2016-03-11 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Alcohol Dependence
Keywords: alcohol use disorders; physical activity; women's health
MeSH Terms: conditions — Alcoholism; Motor Activity

STUDY DESIGN:
Intervention Model Description: RCT

ARMS (2):
- LPA+Fitbit (Experimental): A 12-week LPA+Fitbit intervention for depressed women in intensive alcohol treatment. This will include: 1) a single in-person physical activity (PA) counseling orientation session; 2) 6 brief, phone-based PA counseling sessions focused on increasing PA and strategically using bouts of PA to cope with affect and alcohol cravings; 3) use of the Fitbit fitness tracker for physical activity goal-setting and daily self-monitoring; and 4) weekly supportive messages delivered by email.
  Interventions: Behavioral: LPA+Fitbit
- Health Education Contact Control (HEC) (Active Comparator): The HEC condition will include: 1) an in-person orientation session, 2) 6 telephone-delivered health education sessions, and 3) weekly health-related e-mails. A variety of health and lifestyle topics will be addressed including the following: Session 1 (week 1) - Nutrition-What to Eat and What Not to Eat; Session 2 (week 2) - Sleep Problems and Sleep Hygiene; Session 3 (week 4) - Alcohol Use among Women; Session 4 (week 6) - Relaxation training; Session 5 (week 8) - Time Management and Assertiveness; and Session 6 (week 10) - Being a Smart Patient when Coordinating your Healthcare.
  Interventions: Behavioral: HEC

INTERVENTIONS:
Behavioral: LPA+Fitbit
  Arms: LPA+Fitbit
Behavioral: HEC
  Arms: Health Education Contact Control (HEC)

SUMMARY:
Building on the large body of evidence for the effect of exercise in decreasing depressive symptoms and the few preliminary findings of its effect on craving and drinking outcomes, the purpose of this study is to develop a lifestyle physical activity (LPA) intervention that harnesses the technological advantages of the Fitbit tracker (plus its web and mobile platforms) for depressed women with alcohol use disorders (AUDs). The intervention will provide women with an acceptable, flexible and effective alternate coping strategy during early recovery, when relapse risk is highest. The overall objective of this work is to fully develop this LPA+Fitbit intervention, modify it based on initial piloting and feedback to ensure its feasibility and acceptability for depressed women with AUDs in early recovery, propose potential mechanisms of its effect, and to obtain preliminary data on its efficacy.

DETAILED DESCRIPTION:
Alcohol use disorders (AUDs) are the 3rd leading preventable cause of death in the U.S. and are associated with significant economic burden and health-related negative consequences. While women may be less likely to develop AUDs, they experience more significant negative health consequences of alcohol use than men. Due to stigma, shame, and child care issues; women are less likely to receive specialty addiction treatment. The comorbidity of depression and AUDs is much higher in women, and compared to men, women depression often has a temporal onset prior to an AUD. Relapse rates are very high in both men and women but significant gender differences emerge in the predictors of relapse. Women are more likely to relapse in unpleasant, negative emotional states and depressive symptoms and negative affect mediate the relationship between these stressors and drinking outcomes. More so than men, women with AUDs report drinking to cope with negative emotions. Therefore, intervention approaches that help women develop alternate coping strategies can have an important role in decreasing alcohol relapse among depressed women with AUDs. Given the demonstrated benefits of exercise for decreasing depression, negative affect, and urges to drink, helping women engage in a flexible and acceptable lifestyle physical activity (LPA) intervention may provide them a tool they can utilizing "in the moment" to cope with negative emotional states and alcohol craving during early recovery when relapse risk is highest. Exciting new digital fitness technologies (e.g., Fitbit activity monitor with web and mobile applications) have emerged in recent years that include features able to further enhance critical components for increasing physical activity - goal setting and self-monitoring. The investigators propose to develop a 12-week LPA+Fitbit intervention for depressed women in alcohol treatment. This will include: 1) an in-person physical activity (PA) counseling orientation session; 2) 4 brief, phone-based PA counseling sessions focused on increasing PA and strategically using bouts of PA to cope with affect and alcohol cravings; 3) use of the Fitbit fitness tracker for physical activity goal-setting and daily self-monitoring; and 4) weekly supportive messages delivered by text message. The overall objective of this application is to develop this LPA+Fitbit intervention, modify it based on a initial open pilot (n=20) and feedback to ensure its feasibility and acceptability for depressed women with AUDs in early recovery, propose potential mechanisms, and to obtain preliminary data on its efficacy in a small randomized clinical trial (n=50). The LPA+Fitbit intervention proposed in this application is simple, low-cost, and easily transportable to the varied clinical settings women with AUDs receive treatment. If women with AUDs find the LPA+Fitbit intervention feasible, acceptable, and helpful during early recovery, they could be afforded with a much needed alternate coping strategy that would reduce relapse risk and decrease the overall negative impact of alcohol use on their health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* currently engaged in alcohol treatment
* meets criteria for DSM-5 alcohol use disorder
* score of 1 on ONE of the first 2 items of the Patient Health Questionnaire (PHQ-9)
* less than 150 minutes of moderate-intensity aerobic exercise per week over the last 6 months
* has access to a computer connected to the internet or a smartphone compatible with the Fitbit application

Exclusion Criteria:

* current DSM-5 diagnosis of moderate/severe substance use disorder, anorexia, or bulimia
* history of psychotic disorder or current psychotic symptoms
* current suicidality or homicidality
* current mania
* marked organic impairment
* physical or medical problems that would not allow safe participation in exercise
* currently pregnant or intending to be pregnant in the next 12 weeks

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent | 6-months

SECONDARY OUTCOMES:
Level of depressive symptoms as measured by the Quick Inventory of Depressive Symptomatology (QIDS) | 6-months
Steps/day as measured by the actigraphy | 6-months
Positive coping scores on the Brief COPE measure | 6-months
Level of motivation for abstinence using the Contemplation Ladder | 6-months
Level of self-efficacy on the Alcohol Abstinence Self-Efficacy Scale | 6-months
estimated VO2 max on the 6-minute Astrand-Rhyming Cycle Test | 6-months

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States